CLINICAL TRIAL: NCT05446818
Title: Intra-individual Real Life Effects of Cocoa Flavanols on Blood Pressure and Arterial Stiffness Using Personal Devices in Healthy Humans: Series of Repeated Cross-over Randomized Controlled Double-blind N-of-1 Pilot Studies
Brief Title: Intra-individual Real Life Effects of Cocoa Flavanols on Blood Pressure and Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FER-1819-040
Record Dates: First submitted 2019-04-26; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2021-05

CONDITIONS: Blood Pressure; Stiffness, Vascular; Sleep

STUDY DESIGN:
Intervention Model Description: Series of Repeated Cross-over Randomized Controlled Double-blind N-of-1 Pilot Studies; each subject receives 4 times treatment and 4 times placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Intervention and placebo in same number and size of capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flavanol first (Active Comparator): Subjects will receive over 8 days both cocoa flavanols (CF) and placebo (P) capsules on alternating days. Sequence of this arm is: CF-P-CF-P-CF-P-CF-P
  Interventions: Dietary Supplement: Cocoa flavanol (CF); Other: Placebo (P)
- Placebo first (Active Comparator): Subjects will receive over 8 days both cocoa flavanols (CF) and placebo (P) capsules on alternating days. Sequence of this arm is: P-CF-P-CF-P-CF-P-CF
  Interventions: Dietary Supplement: Cocoa flavanol (CF); Other: Placebo (P)

INTERVENTIONS:
Dietary Supplement: Cocoa flavanol (CF) — 2 times per day 750 mg cocoa flavanols (each delivered in 6 CocoaVia capsules)
Other: Placebo (P) — 2 times per day 0 mg cocoa flavanols calorically matched control (delivered in 6 identical capsules)

SUMMARY:
Very controlled dietary intervention studies support that individual polyphenol rich foods and isolated polyphenols can increase endothelial function and HDL cholesterol and decrease blood pressure, arterial stiffness, and LDL cholesterol even in healthy subjects. The intake of (-)-epicatechin, the major polyphenol in cocoa, was previously mechanistically linked with acute improvements in endothelial function and nitric oxide availability. A profound understanding of inter- and intra-individual variability of responses in real life are an important area of research in a world that aims at personalized nutrition and medicine. N-of-1 trials are a powerful tool allowing to study small effects even in fewer subjects and help account for intra-individual variations in responses. The overall aim of the present pilot study is to evaluate intra-and inter-individual variability of responses to cocoa flavanols in everyday life using the N-of-1 paradigm. In this pilot study, young healthy humans will monitor blood pressure, pulse wave velocity, heart rate, diet, and physical activity on 8 days using a personal and wearable devices. Each subject will undergo the 8 study days; 4 days with cocoa flavanol capsules (CF; containing 750 mg (1500 mg per day)) and 4 days with calorically matched placebo capsules (P; 0 mg cocoa flavanols) taken at the same time in the morning with breakfast and at night before going to bed. The subjects will be randomized to different treatment allocation sequences to allow blinding of volunteers and investigator; either CF-P-CF-P-CF-P-CF-P or P-CF-P-CF-P-CF-P-CF.

DETAILED DESCRIPTION:
Background: Very controlled dietary intervention studies support that individual polyphenol rich foods and isolated polyphenols can increase endothelial function and HDL cholesterol and decrease blood pressure, arterial stiffness, and LDL cholesterol even in healthy subjects. The intake of (-)-epicatechin, the major polyphenol in cocoa, was previously mechanistically linked with acute improvements in endothelial function and nitric oxide availability. However, the clinical intervention studies were performed in tightly controlled experimental settings and variability of individual responses were not investigated. A profound understanding of inter- and intra-individual variability of responses in real life are an important area of research in a world that aims at personalized nutrition and medicine. N-of-1 trials are a powerful tool allowing to study small effects even in fewer subjects and help account for intra-individual variations in responses. N-of-1 trials in clinical medicine are multiple crossover trials, usually randomized and often blinded, conducted in a single patient.

Aim, hypothesis, objectives: The overall aim of the present pilot study is to evaluate intra-and inter-individual variability of responses to cocoa flavanols in everyday life using the N-of-1 paradigm. It is the hypothesis that cocoa flavanols decrease blood pressure and arterial stiffness in everyday life of healthy individuals. The objectives to investigate the aim are (1) to test the effect of CF using wearable devices repeatedly measuring blood pressure, arterial stiffness, and heart rate in healthy individuals participating in in every days life, (2) to explore intra-and inter-individual variability in responses by repeatedly testing responses in the same individuals, and (3) to test different statistical models taking repeated measurements in the same subject into account.

Methods: In this pilot study, young healthy humans will monitor blood pressure, pulse wave velocity, heart rate, diet, and physical activity on 8 days using a personal and wearable devices. Each subject will undergo the 8 study days; 4 days with cocoa flavanol capsules (CF; containing 750 mg (1500 mg per day)) and 4 days with calorically matched placebo capsules (P; 0 mg cocoa flavanols) taken at the same time in the morning with breakfast and at night before going to bed. The subjects will be randomized to different treatment allocation sequences to allow blinding of volunteers and investigator; either CF-P-CF-P-CF-P-CF-P or P-CF-P-CF-P-CF-P-CF. Blood pressure and heart rate will be measured by a standard upper arm blood pressure cuff and estimated by a fitness wristband and pulse wave velocity via a finger device in 30 min intervals for 3 h starting after morning treatment ingestion followed by hourly intervals until going to bed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body mass index <30 kg/m2
* Age <45 years

Exclusion Criteria:

* Diabetes mellitus
* Symptoms of acute infection
* Cardiac arrhythmia
* Active malignancy
* Clinical signs or symptoms of cardiovascular disease including:

  1. Angina pectoris
  2. Shortness of breath
  3. Palpitations
  4. Syncopes
  5. Claudication
* Active vasoactive medication
* Vitamin supplements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Measurements over 24 hours
  Standard upper arm cuff (day) and wrist band (day and night)
Change in arterial stiffness | Measurements over 24 hours
  Pulse wave velocity by finger clip (iHeart)
Change in heart rate | Measurements over 24 hours
  Fitness bracelet

SECONDARY OUTCOMES:
Physical activity | Assessed over 24 hours
  Steps measured on fitness bracelet

OTHER OUTCOMES:
Dietary composition | Assessed over 24 hours
  Dietary assessment based on food diary

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No